CLINICAL TRIAL: NCT02925819
Title: Management And Clinical Outcomes Of Patients With Severe Mitral Disease Not Suitable For Surgery: A Prospective, Multicentric, Observational Study
Brief Title: Management and Clinical Outcomes of Patients With Severe Mitral Valve Disease Not Suitable for Surgery
Acronym: MITRAGISTER
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 15.534
Record Dates: First submitted 2016-09-08; First posted 2016-10-06 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mitral Valve Disease
Keywords: Mitral regurgitation; Mitral stenosis; Mitral valve repair deterioration; Bioprosthesis degeneration
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SEVERE MITRAL VALVE DISEASE: All patients with symptomatic severe mitral valve disease on a native valve or due to deterioration after surgical valve repair or replacement, and not eligible for surgery according to the heart-team.

SUMMARY:
The objective of this study is to collect in a prospective registry all cases of French patients undergoing an assessment for percutaneous treatment of mitral valve disease on a native valve or due to deterioration after surgical valve repair or replacement. In these patients, valvular surgery should be considered contra-indicated or at prohibitive risk. This registry will evaluate the morbidity and mortality up to 24 months for those patients with severe mitral valve disease who are not included in a clinical trial. The association of demographic, clinical, laboratory, echocardiographic variables and treatment options with morbidity and mortality will be evaluated by univariate and multivariate analyses.

DETAILED DESCRIPTION:
Patients with symptomatic severe mitral valve disease will have a medical evaluation visit (physical examination, ECG, biology) with transthoracic ± transesophageal echocardiography in each center. If the patient is considered not eligible for surgery by the heart-team and is not included in a clinical trial, the investigator informs the patient of the existence of the registry and verifies that it does not express opposition to the use of its clinical data.

In each participating center, demographic information, clinical, laboratory, echocardiographic and treatment options will be collected and reported in an electronic case report form (e-CRF). Each center will be responsible of patient monitoring, including phone call at 6 months and a medical visit at 1 and 2 years. Transthoracic echocardiography will also be performed at 1 year and 2 years.

ELIGIBILITY:
* Aged over 18 years
* Presenting with severe mitral valve stenosis or regurgitation regardless of etiology (primary mitral regurgitation, secondary mitral regurgitation, deterioration of mitral valve repair or bioprosthesis, mitral annular calcification)
* Symptomatic (NYHA functional class II-IV) despite optimized medical therapy
* Judged not eligible for surgical treatment according to a specialized multidisciplinary meeting called "heart team" comprising at least one cardiothoracic surgeon, one interventional cardiologist, one echocardiographer, one clinical cardiologist and one anaesthesiologist.
* Having received information about the study and not expressing opposition to the use of their data
* Patient not included in a clinical trial

Exclusion Criteria:

* Asymptomatic patients
* Absence of severe mitral regurgitation or stenosis
* Patient judged eligible for surgical treatment according to a specialized multidisciplinary meeting called "heart team" comprising at least one cardiothoracic surgeon, one interventional cardiologist, one echocardiographer, one clinical cardiologist and one anaesthesiologist.
* Pregnant or breastfeeding women
* Having not received information about the study or having expressed opposition to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients undergoing an assessment for percutaneous treatment of symptomatic severe mitral valve disease on a native valve or due to deterioration after surgical valve repair or replacement with contra-indication to or prohibitive risk of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All cause death and heart failure at 24 months | 24 months of follow-up
  Death from any cause or unscheduled hospitalization for heart failure at 24 months

SECONDARY OUTCOMES:
Overall survival at 24 months | 24 months of follow-up
  The survival rate will be determined between the date of inclusion in the cohort and the date of occurrence of death, whatever the cause.
Survival without major cardiovascular event | 24 months of follow-up
  The rate of survival without major cardiovascular event rate will be determined between the date of inclusion and date of occurrence of a major cardiovascular event (unscheduled rehospitalisation for heart failure, stroke, death of cardiovascular, myocardial infarction).
Rate of unscheduled hospitalizations for heart failure | 24 months of follow-up
  Rate of unscheduled hospitalizations for heart failure at 24 months.
Functional evaluation | 24 months of follow-up
  It will be defined by changes in NYHA functional class at 24 months.
Early safety | Until Hospital Discharge, up to 6 months
  Defined as absence of all-cause mortality, all stroke, severe bleeding, acute kidney injury stage 2 or 3, major vascular complication, and valve related dysfunction requiring repeat interventional transcatheter procedure or surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François OBADIA, Principal Investigator — Hospices Civils de Lyon; Bernard IUNG, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Patrice GUERIN, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - CHU Lyon, Lyon
  - CHU Nantes, Nantes
  - Bichat Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698
- [Background] De Bonis M, Lapenna E, La Canna G, Ficarra E, Pagliaro M, Torracca L, Maisano F, Alfieri O. Mitral valve repair for functional mitral regurgitation in end-stage dilated cardiomyopathy: role of the "edge-to-edge" technique. Circulation. 2005 Aug 30;112(9 Suppl):I402-8. doi: 10.1161/CIRCULATIONAHA.104.525188. PMID 16159854
- [Background] Alfieri O, Maisano F, De Bonis M, Stefano PL, Torracca L, Oppizzi M, La Canna G. The double-orifice technique in mitral valve repair: a simple solution for complex problems. J Thorac Cardiovasc Surg. 2001 Oct;122(4):674-81. doi: 10.1067/mtc.2001.117277. PMID 11581597
- [Background] Whitlow PL, Feldman T, Pedersen WR, Lim DS, Kipperman R, Smalling R, Bajwa T, Herrmann HC, Lasala J, Maddux JT, Tuzcu M, Kapadia S, Trento A, Siegel RJ, Foster E, Glower D, Mauri L, Kar S; EVEREST II Investigators. Acute and 12-month results with catheter-based mitral valve leaflet repair: the EVEREST II (Endovascular Valve Edge-to-Edge Repair) High Risk Study. J Am Coll Cardiol. 2012 Jan 10;59(2):130-9. doi: 10.1016/j.jacc.2011.08.067. PMID 22222076
- [Background] Maisano F, Franzen O, Baldus S, Schafer U, Hausleiter J, Butter C, Ussia GP, Sievert H, Richardt G, Widder JD, Moccetti T, Schillinger W. Percutaneous mitral valve interventions in the real world: early and 1-year results from the ACCESS-EU, a prospective, multicenter, nonrandomized post-approval study of the MitraClip therapy in Europe. J Am Coll Cardiol. 2013 Sep 17;62(12):1052-1061. doi: 10.1016/j.jacc.2013.02.094. Epub 2013 Jun 7. PMID 23747789
- [Background] Baldus S, Schillinger W, Franzen O, Bekeredjian R, Sievert H, Schofer J, Kuck KH, Konorza T, Mollmann H, Hehrlein C, Ouarrak T, Senges J, Meinertz T; German Transcatheter Mitral Valve Interventions (TRAMI) investigators. MitraClip therapy in daily clinical practice: initial results from the German transcatheter mitral valve interventions (TRAMI) registry. Eur J Heart Fail. 2012 Sep;14(9):1050-5. doi: 10.1093/eurjhf/hfs079. Epub 2012 Jun 8. PMID 22685268
- [Background] Armoiry X, Brochet E, Lefevre T, Guerin P, Dumonteil N, Himbert D, Cormier B, Piriou N, Gautier M, Messika-Zeitoun D, Romano M, Rioufol G, Warin Fresse K, Boudou N, Leclercq F, Bedossa M, Obadia JF. Initial French experience of percutaneous mitral valve repair with the MitraClip: a multicentre national registry. Arch Cardiovasc Dis. 2013 May;106(5):287-94. doi: 10.1016/j.acvd.2013.03.059. Epub 2013 May 28. PMID 23769403
- [Background] Obadia JF, Armoiry X, Iung B, Lefevre T, Mewton N, Messika-Zeitoun D, Cormier B, Berthiller J, Maucort-Boulch D, Boutitie F, Vaz B, Trochu JN, Vahanian A. The MITRA-FR study: design and rationale of a randomised study of percutaneous mitral valve repair compared with optimal medical management alone for severe secondary mitral regurgitation. EuroIntervention. 2015 Mar;10(11):1354-60. doi: 10.4244/EIJV10I11A232. PMID 25798568